CLINICAL TRIAL: NCT00333866
Title: A 14 Week, Randomized, Double-Blind, Placebo-Controlled Trial Of Pregabalin Twice Daily In Patients With Fibromyalgia.
Brief Title: Randomized, Double-Blind, Placebo-Controlled Trial Of Pregabalin In Patients With Fibromyalgia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081100
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2009-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: pregabalin
- 2 (Experimental)
  Interventions: Drug: pregabalin
- 3 (Experimental)
  Interventions: Drug: pregabalin
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — 600mg/day
  Arms: 1
Drug: pregabalin — 450mg/day
  Arms: 2
Drug: pregabalin — 300mg/day
  Arms: 3
Drug: placebo — placebo
  Arms: 4

SUMMARY:
This study, will compare pregabalin with placebo for the duration of 14 weeks to evaluate the efficacy and safety of pregabalin in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria for fibromyalgia
* A score of more or equal to 40 mm on the Pain Visual Analog Scale (VAS) and a an average score more or equal to 4 on 4 daily pain diaries

Exclusion Criteria:

* Patients with other severe pain conditions
* Patients with severe depression
* Patients taking excluded medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- Australia (4):
  - Pfizer Investigational Site, Warrawong, New South Wales
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Fitzroy, Victoria
- Canada (11):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Denmark (2):
  - Pfizer Investigational Site, Frederiksberg
  - Pfizer Investigational Site, Svendborg
- France (5):
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Lille, Cedex
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Etienne
- Germany (5):
  - Pfizer Investigational Site, Bad Säckingen
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
- India (3):
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Italy (6):
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Benevento
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Chieti Scalo
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
- Mexico (4):
  - Pfizer Investigational Site, México, D. F.
  - Pfizer Investigational Site, León, Guanajuato
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, San Luis Potosí City
- Netherlands (5):
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Den Helder
  - Pfizer Investigational Site, Leeuwarden
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Zwolle
- Pfizer Investigational Site, Lisbon, Portugal
- South Korea (2):
  - Pfizer Investigational Site, Suwon, Kyeongki-do
  - Pfizer Investigational Site, Seoul
- Spain (3):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Córdoba
  - Pfizer Investigational Site, Guadalajara
- Sweden (4):
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
- Switzerland (2):
  - Pfizer Investigational Site, Lausanne
  - Pfizer Investigational Site, Zurich
- United Kingdom (5):
  - Pfizer Investigational Site, Manchester, Greater Manchester
  - Pfizer Investigational Site, Greenock, Renfrewshire
  - Pfizer Investigational Site, North Shields, Tyne and Wear
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Poole
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, Distrito Federal
  - Pfizer Investigational Site, Caracas, Miranda

REFERENCES:
- [Derived] Clair A, Emir B. The safety and efficacy of pregabalin for treating subjects with fibromyalgia and moderate or severe baseline widespread pain. Curr Med Res Opin. 2016;32(3):601-9. doi: 10.1185/03007995.2015.1134463. Epub 2016 Jan 27. PMID 26694975
- [Derived] Pauer L, Winkelmann A, Arsenault P, Jespersen A, Whelan L, Atkinson G, Leon T, Zeiher B; A0081100 Investigators. An international, randomized, double-blind, placebo-controlled, phase III trial of pregabalin monotherapy in treatment of patients with fibromyalgia. J Rheumatol. 2011 Dec;38(12):2643-52. doi: 10.3899/jrheum.110569. Epub 2011 Oct 1. PMID 21965636
- [Derived] Straube S, Moore RA, Paine J, Derry S, Phillips CJ, Hallier E, McQuay HJ. Interference with work in fibromyalgia: effect of treatment with pregabalin and relation to pain response. BMC Musculoskelet Disord. 2011 Jun 3;12:125. doi: 10.1186/1471-2474-12-125. PMID 21639874
- [Derived] Bhadra P, Petersel D. Medical conditions in fibromyalgia patients and their relationship to pregabalin efficacy: pooled analysis of Phase III clinical trials. Expert Opin Pharmacother. 2010 Dec;11(17):2805-12. doi: 10.1517/14656566.2010.525217. Epub 2010 Nov 2. PMID 21039311
- [Derived] Bennett RM, Russell J, Cappelleri JC, Bushmakin AG, Zlateva G, Sadosky A. Identification of symptom and functional domains that fibromyalgia patients would like to see improved: a cluster analysis. BMC Musculoskelet Disord. 2010 Jun 28;11:134. doi: 10.1186/1471-2474-11-134. PMID 20584327
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081100&StudyName=Randomized%2C%20Double-Blind%2C%20Placebo-Controlled%20Trial%20Of%20Pregabalin%20%20In%20Patients%20With%20Fibromyalgia.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 73 centers in North America [Canada (12) and Mexico (4)], South America [Venezuela (3)], Europe [Denmark (2), France (5), Germany (5), Italy (6), Netherlands (5), Portugal (4), Spain (4), Sweden (4), Switzerland (3) and United Kingdom(5)] and Asia [India (4) and Korea (3)] and Australia (4).
Groups:
- Placebo: Placebo matched to pregabalin capsules orally twice daily up to Week 14.
- Pregabalin 300 mg: Pregabalin capsule 150 milligram (mg) orally twice daily following a 2 week titration phase, Day 1-3: 75 mg orally twice daily and Day 4 onwards: 150 mg orally twice daily fixed dose up to Week 14.
- Pregabalin 450 mg: Pregabalin capsule 225 mg orally twice daily following a 2 week titration phase, Day 1-3: 75 mg orally twice daily, Day 4-8: 150 mg orally twice daily, Day 9-11: 200 mg orally twice daily and Day 12 onwards: 225 mg orally twice daily fixed dose up to Week 14.
- Pregabalin 600 mg: Pregabalin capsule 300 mg orally twice daily following a 2 week titration phase, Day 1-3: 75 mg orally twice daily, Day 4-8: 150 mg orally twice daily, Day 9-11: 200 mg orally twice daily and Day 12-14: 225 mg orally twice daily and then 300 mg orally twice daily fixed dose up to Week 14.
Period: Overall Study
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Started | 189 | 187 | 184 | 187
TREATED | 184 | 184 | 182 | 186
Completed | 141 | 123 | 133 | 121
Not Completed | 48 | 64 | 51 | 66
Not completed — Adverse Event | 23 | 37 | 38 | 47
Not completed — Other | 3 | 2 | 2 | 2
Not completed — Lack of Efficacy | 8 | 6 | 3 | 5
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 8 | 14 | 4 | 9
Not completed — Randomized but not Treated | 5 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg | Total
Number analyzed (Participants) | 184 | 184 | 182 | 186 | 736
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.3) | 48.4 (10.8) | 48.0 (11.3) | 49.6 (11.3) | 48.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 167 | 169 | 169 | 673
  Male | 16 | 17 | 13 | 17 | 63
Mean Pain Score [Mean (Standard Deviation); unit: Units on a scale] — Daily pain diary consists of 11-point numeric rating scale (NRS) ranging from 0(no pain) to 10(worst possible pain). Participants rated their pain during past 24 hours, self-assessment done daily at awakening. Baseline=Last 7 available pain scores before taking study medication up to and including Day 1. Number of participants evaluable=184,184,181,186.
  Units on a scale | 6.68 (1.48) | 6.76 (1.29) | 6.57 (1.31) | 6.59 (1.37) | 6.65 (1.36)
Mean Sleep Quality Score [Mean (Standard Deviation); unit: Units on a scale] — Daily quality of sleep diary consists of 11-point NRS ranging from 0(best possible sleep) to 10(worst possible sleep). Participants rated their quality of sleep during past 24 hours, self-assessment done daily upon awakening. Baseline=Last 7 available scores before taking study medication up to and including Day 1. Number of participants evaluable=184,184,181,186.
  Units on a scale | 6.01 (1.90) | 5.94 (1.70) | 5.94 (1.70) | 5.91 (1.80) | 5.95 (1.77)
Percentage of Participants With Optimal Sleep Assessed Using MOS-SS [Number; unit: Percentage of Participants] — MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Percentage of participants with optimal sleep are reported. Number of participants evaluable=182,182,175,182.
  Percentage of Participants | 20.33 | 25.27 | 24.57 | 17.03 | 87.2
Medical Outcome Study Sleep Scale (MOS-SS) [Mean (Standard Deviation); unit: Units on a scale] — Participant-rated 12 item questionnaire assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no), as well as a 9-item overall sleep problems index. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score minus lowest possible score divided by possible raw score range*100);total score range:0-100,higher score=more intensity of attribute. Number of participants evaluable=183,183,177,185.
  Units on a scale
    Sleep Disturbance | 60.02 (25.60) | 61.86 (25.80) | 59.59 (26.55) | 60.37 (25.09) | 60.47 (25.72)
    Snoring | 31.05 (32.39) | 32.53 (30.82) | 29.77 (32.52) | 32.09 (32.20) | 31.36 (31.94)
    Shortness of Breath, Headache | 34.18 (32.96) | 36.70 (31.01) | 38.31 (32.46) | 37.07 (31.54) | 36.55 (31.97)
    Quantity of Sleep | 5.47 (1.54) | 5.59 (1.66) | 5.61 (1.68) | 5.45 (1.65) | 5.53 (1.63)
    Sleep Adequacy | 24.70 (23.39) | 24.43 (24.80) | 24.30 (22.83) | 25.03 (24.25) | 24.62 (23.79)
    Somnolence | 41.68 (21.78) | 44.03 (22.80) | 42.37 (23.91) | 42.97 (23.92) | 42.77 (23.09)
    Overall Sleep Problem Index | 57.46 (17.27) | 59.27 (19.24) | 58.11 (18.94) | 58.05 (18.12) | 58.22 (18.38)
Fibromyalgia Impact Questionnaire (FIQ) Subscale Scores [Mean (Standard Deviation); unit: Units on a scale] — FIQ: 20-item self-administered questionnaire designed to assess areas such as health status, progress, and outcomes in participants with fibromyalgia. 11 items related to physical functioning, other items assess pain, fatigue, stiffness, difficulty working, and symptoms of anxiousness and depression. FIQ contains 10 sub-scales scored from 0 to 10, with higher scores indicating more impairment in the subscale attribute. Total score range from 0 to 100 with higher scores indicating more impairment. Number of participants evaluable=183,184,179,186.
  Units on a scale
    FIQ Physical Impairment | 4.04 (2.18) | 3.88 (2.13) | 3.87 (2.12) | 3.75 (2.15) | 3.88 (2.14)
    FIQ Feel Good | 7.50 (2.61) | 7.46 (2.77) | 7.63 (2.53) | 7.77 (2.65) | 7.59 (2.64)
    FIQ Work Missed | 3.38 (3.34) | 3.35 (3.18) | 3.22 (3.36) | 2.86 (2.99) | 3.20 (3.22)
    FIQ Do Work | 6.96 (2.24) | 6.54 (2.23) | 6.68 (1.96) | 6.62 (2.01) | 6.70 (2.12)
    FIQ Pain | 7.35 (1.63) | 7.24 (1.48) | 7.09 (1.62) | 7.15 (1.60) | 7.21 (1.58)
    FIQ Fatigue | 7.85 (1.84) | 7.45 (2.14) | 7.34 (2.02) | 7.56 (2.04) | 7.55 (2.02)
    FIQ Rested | 7.71 (2.03) | 7.61 (2.08) | 7.55 (1.96) | 7.44 (2.02) | 7.58 (2.02)
    FIQ Stiffness | 7.52 (2.13) | 7.19 (2.07) | 7.03 (2.02) | 7.28 (2.24) | 7.26 (2.12)
    FIQ Anxiety | 5.38 (3.09) | 5.27 (2.96) | 5.35 (2.86) | 5.35 (2.97) | 5.34 (2.97)
    FIQ Depression | 4.85 (3.12) | 4.73 (2.93) | 4.79 (3.01) | 4.65 (3.00) | 4.76 (3.01)
Fibromyalgia Impact Questionnaire (FIQ) Total Scores [Mean (Standard Deviation); unit: Units on a scale] — FIQ: 20-item self-administered questionnaire designed to assess areas such as health status, progress, and outcomes in participants with fibromyalgia. 11 items related to physical functioning, other items assess pain, fatigue, stiffness, difficulty working, and symptoms of anxiousness and depression. FIQ contains 10 sub-scales scored from 0 to 10, with higher scores indicating more impairment in the subscale attribute. Total score range from 0 to 100 with higher scores indicating more impairment. Number of participants evaluable=184,184,179,186.
  Units on a scale | 62.58 (14.85) | 60.75 (14.77) | 60.59 (14.59) | 60.40 (13.87) | 61.08 (14.52)
36-Item Short-Form Health Survey (SF-36) [Mean (Standard Deviation); unit: Units on a scale] — SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; Physical Component Score and Mental Component Score. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning. Number of participants evaluable=184,184,181,186.
  Units on a scale
    Physical Functioning | 42.93 (21.04) | 44.71 (20.29) | 42.52 (22.17) | 43.54 (20.39) | 43.43 (20.94)
    Physical Role Limitations | 37.14 (22.75) | 40.79 (25.58) | 41.44 (25.39) | 39.46 (24.71) | 39.69 (24.63)
    Emotional Role Limitations | 59.61 (29.52) | 60.61 (29.23) | 61.54 (28.94) | 61.31 (29.50) | 60.76 (29.25)
    Social Functioning | 54.44 (26.95) | 56.79 (26.00) | 53.93 (26.55) | 53.70 (25.55) | 54.72 (26.24)
    Mental Health | 56.48 (20.68) | 56.41 (20.49) | 57.56 (21.70) | 56.71 (20.39) | 56.78 (20.77)
    Bodily Pain | 29.28 (15.61) | 28.67 (13.65) | 28.30 (13.62) | 28.70 (13.20) | 28.74 (14.03)
    Vitality | 26.46 (16.76) | 27.88 (17.67) | 28.78 (19.94) | 27.42 (19.14) | 27.63 (18.39)
    General Health Perception | 41.65 (18.35) | 42.12 (19.24) | 45.56 (18.56) | 44.58 (18.23) | 43.47 (18.63)
    Mental Component Score | 40.11 (11.57) | 40.45 (11.72) | 40.79 (13.15) | 40.37 (12.14) | 40.43 (12.13)
    Physical Component Score | 31.87 (7.59) | 32.60 (7.43) | 32.51 (8.16) | 32.42 (7.03) | 32.35 (7.55)
Multidimensional Assessment of Fatigue (MAF) [Mean (Standard Deviation); unit: Units on a scale] — MAF is a 16-item self-administered questionnaire that yields a Global Fatigue Index (GFI), measures 4 dimensions of fatigue: degree and severity, amount of distress it causes, its timing and degree to which fatigue interferes with activities of daily living. Only 15 items are used to calculate the GFI. GFI score range from 1 (no fatigue) to 50 (severe fatigue). Number of participants evaluable=183,176,175,181.
  Units on a scale | 34.89 (7.52) | 34.97 (7.71) | 33.98 (8.29) | 34.87 (7.70) | 34.68 (7.80)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: Units on a scale] — HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms. Number of participants evaluable=182,181,176,185.
  Units on a scale
    HADS Anxiety (HADS-A) Total | 8.95 (4.52) | 8.96 (4.50) | 8.75 (4.44) | 8.85 (4.58) | 8.88 (4.51)
    HADS Depression (HADS-D) Total | 7.83 (4.17) | 7.16 (4.03) | 7.66 (4.32) | 7.39 (4.28) | 7.51 (4.20)
Pain Visual Analogue Scale (VAS) Scores [Mean (Standard Deviation); unit: millimeter (mm)] — Pain visual analog scale (VAS): Participants assessed the severity of their pain using a 100 mm visual analog scale (VAS). The scale ranged from 0 (no pain) to 100 (worst possible pain), measurement on a scale corresponds to the magnitude of their pain. Number of participants evaluable=184,184,181,186.
  millimeter (mm) | 72.72 (14.09) | 72.43 (13.61) | 70.92 (13.69) | 71.43 (13.51) | 71.88 (13.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Pain Score at Endpoint (Up to Week 14)
Description: Daily pain diary consists of 11-point NRS ranging from 0(no pain) to 10(worst possible pain). Participants rated their pain during past 24 hours, self-assessment done daily at awakening. Baseline=Last 7 available pain scores before taking study medication up to and including Day 1. Final weekly (endpoint) mean pain score is defined as the mean pain score from the last 7 pain diary entries in the study while the participant was on study medication.
Time Frame: Baseline, Week 14
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. Missing data were imputed using last observation carried forward (LOCF) method. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 181 | 186
Units on a scale | -0.73 (0.14) | -1.06 (0.14) | -1.29 (0.14) | -0.96 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P value was calculated using Analysis of Covariance (ANCOVA) with treatment and center in the model, and the baseline mean pain score as covariate; Test type: Superiority or Other; p = 0.2361, ANCOVA; Hochberg's approach was used to protect the Type I error rate at 0.05 level, Hochberg adjusted p-values were presented; Least Squares (LS) mean difference = -0.23, 95% CI 2-sided [-0.61 to 0.15]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; P value was calculated using ANCOVA with treatment and center in the model, and the baseline mean pain score as covariate; Test type: Superiority or Other; p = 0.0132, ANCOVA; Hochberg's approach was used to protect the Type I error rate at 0.05 level, Hochberg adjusted p-values were presented; LS mean difference = -0.56, 95% CI 2-sided [-0.94 to -0.17]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1694, ANCOVA; Hochberg's approach was used to protect the Type I error rate at 0.05 level, Hochberg adjusted p-values were presented; Least Squares (LS) mean difference = -0.33, 95% CI 2-sided [-0.72 to 0.05]

2. Primary Outcome: Patient Global Impression of Change (PGIC)
Description: Number of participants with categorical change in overall status. PGIC: a participant-rated instrument assessing change in participant's overall status from baseline, on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 14
Population: FAS included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. Missing data were imputed using LOCF method. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 169 | 164 | 165 | 155
participants
  Very much improved | 7 | 13 | 16 | 20
  Much improved | 43 | 45 | 50 | 46
  Minimally improved | 45 | 50 | 55 | 41
  No change | 43 | 28 | 27 | 25
  Minimally worse | 11 | 9 | 7 | 10
  Much worse | 17 | 14 | 8 | 10
  Very much worse | 3 | 5 | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P-values less than 0.05 (2-sided) considered statistically significant. P-values were calculated using a modified ridit transformation with the Cochran-Mantel-Haenszel procedure, adjusting for center; Test type: Superiority or Other; p = 0.0227, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0768, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Mean Sleep Quality Score at Endpoint (Up to Week 14)
Description: Daily quality of sleep diary consists of 11-point NRS ranging from 0(best possible sleep) to 10(worst possible sleep). Participants rated their quality of sleep during past 24 hours, self-assessment done daily upon awakening. Baseline=Last 7 available scores before taking study medication up to and including Day 1. The endpoint (up to week 14) mean quality of sleep score was based on Least Squares (LS) Means using ANCOVA, with treatment group and center in the model and the baseline mean sleep score used as the covariate. Final weekly (endpoint) mean sleep quality score is defined as the mean sleep quality score from the last 7 sleep diary entries in the study while the participant was on study medication.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 181 | 186
Units on a scale | -0.94 (0.15) | -1.42 (0.15) | -1.72 (0.15) | -1.95 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline mean sleep score as covariate; Test type: Superiority or Other; p < .0001, ANCOVA; LS mean difference = -1.01, 95% CI 2-sided [-1.42 to -0.60]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; LS mean difference = -0.78, 95% CI 2-sided [-1.20 to -0.37]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0222, ANCOVA; LS mean difference = -0.48, 95% CI 2-sided [-0.89 to -0.07]

4. Secondary Outcome: Change From Baseline in Weekly Mean Sleep Quality Score
Description: Daily quality of sleep diary consists of 11-point NRS ranging from 0(best possible sleep) to 10(worst possible sleep). Participants rated their quality of sleep during past 24 hours, self-assessment done daily upon awakening. Baseline=Last 7 available scores before taking study medication up to and including Day 1. The weekly mean quality of sleep score was based on LS Means using mixed model repeated measures ANCOVA, with treatment, center, week, and treatment-by-week interaction in the model and the baseline mean sleep score used as the covariate. Weekly mean sleep quality score is defined as the mean of the last 7 daily sleep diary entries.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: FAS included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n' participants evaluable at given time point for each group, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 183 | 179 | 174 | 178
Units on a scale
  Week 1 (n=183,179,174,178) | -0.38 (0.14) | -1.20 (0.15) | -1.08 (0.15) | -1.23 (0.15)
  Week 2 (n=180,172,168,174) | -0.62 (0.14) | -1.48 (0.15) | -1.43 (0.15) | -1.59 (0.15)
  Week 3 (n=174, 164, 159,163) | -0.75 (0.15) | -1.42 (0.15) | -1.56 (0.15) | -1.90 (0.15)
  Week 4 (n=165,157,155,156) | -0.73 (0.15) | -1.52 (0.15) | -1.67 (0.15) | -2.01 (0.15)
  Week 5 (n=163, 150, 152,148) | -0.82 (0.15) | -1.67 (0.15) | -1.69 (0.15) | -1.99 (0.15)
  Week 6 (n=159,145,148,144) | -0.84 (0.15) | -1.56 (0.15) | -1.76 (0.16) | -2.15 (0.16)
  Week 7 (n=155,140,144,133) | -0.91 (0.15) | -1.50 (0.16) | -1.83 (0.16) | -2.20 (0.16)
  Week 8 (n=149,133,142,127) | -0.99 (0.15) | -1.60 (0.16) | -1.95 (0.16) | -2.25 (0.16)
  Week 9 (n=146,128,141,126) | -1.11 (0.15) | -1.64 (0.16) | -1.94 (0.16) | -2.24 (0.16)
  Week 10 (n=144,125,139,126) | -1.14 (0.16) | -1.75 (0.16) | -2.03 (0.16) | -2.34 (0.17)
  Week 11 (n=143,123,137,121) | -1.09 (0.16) | -1.65 (0.17) | -1.92 (0.16) | -2.24 (0.17)
  Week 12 (n=141,121,135,119) | -1.22 (0.16) | -1.62 (0.17) | -1.95 (0.16) | -2.29 (0.17)
  Week 13 (n=140,120,133,118) | -1.05 (0.16) | -1.66 (0.17) | -1.93 (0.17) | -2.26 (0.17)
  Week 14 (n=134,115,128,111) | -1.08 (0.16) | -1.73 (0.17) | -1.95 (0.17) | -2.29 (0.18)
  Overall (n=183,179,174,178) | -0.91 (0.12) | -1.57 (0.12) | -1.76 (0.12) | -2.07 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; Week 1: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.85, 95% CI 2-sided [-1.2 to -0.5]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.70, 95% CI 2-sided [-1.1 to -0.3]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.81, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 600 mg; Week 2: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.97, 95% CI 2-sided [-1.3 to -0.6]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.81, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.86, 95% CI 2-sided [-1.2 to -0.5]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 600 mg; Week 3: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.15, 95% CI 2-sided [-1.5 to -0.8]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.80, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.0005, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.67, 95% CI 2-sided [-1.0 to -0.3]
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 600 mg; Week 4: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.28, 95% CI [-1.7 to -0.9]
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.94, 95% CI 2-sided [-1.3 to -0.6]
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.80, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 600 mg; Week 5: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.17, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.87, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.85, 95% CI 2-sided [-1.2 to -0.5]
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 600 mg; Week 6: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.31, 95% CI 2-sided [-1.7 to -0.9]
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.92, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.0003, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.72, 95% CI 2-sided [-1.1 to -0.3]
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 600 mg; Week 7: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.29, 95% CI 2-sided [-1.7 to -0.9]
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.92, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p = 0.0037, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.59, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 600 mg; Week 8: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.27, 95% CI 2-sided [-1.7 to -0.9]
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.97, 95% CI 2-sided [-1.4 to -0.6]
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.0031, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.61, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 600 mg; Week 9: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.12, 95% CI 2-sided [-1.5 to -0.7]
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.83, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p = 0.0117, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.53, 95% CI 2-sided [-0.9 to -0.1]
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 600 mg; Week 10: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.20, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.90, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; p = 0.0040, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.61, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 31: Comparison: Placebo vs Pregabalin 600 mg; Week 11: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.15, 95% CI 2-sided [-1.6 to -0.7]
Statistical Analysis 32: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.83, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 33: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; p = 0.0100, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.56, 95% CI 2-sided [-1.0 to -0.1]
Statistical Analysis 34: Comparison: Placebo vs Pregabalin 600 mg; Week 12: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.07, 95% CI 2-sided [-1.5 to -0.6]
Statistical Analysis 35: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; p = 0.0006, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.73, 95% CI 2-sided [-1.2 to -0.3]
Statistical Analysis 36: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; p = 0.0690, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.40, 95% CI 2-sided [-0.8 to 0.0]
Statistical Analysis 37: Comparison: Placebo vs Pregabalin 600 mg; Week 13: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.21, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 38: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.88, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 39: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; p = 0.0054, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.61, 95% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 40: Comparison: Placebo vs Pregabalin 600 mg; Week 14: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.21, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 41: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 40]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.87, 95% CI 2-sided [-1.3 to -0.4]
Statistical Analysis 42: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 40]; Test type: Superiority or Other; p = 0.0036, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.65, 95% CI 2-sided [-1.1 to -0.2]
Statistical Analysis 43: Comparison: Placebo vs Pregabalin 600 mg; Overall: P-values less than 0.05 (2-sided) considered statistically significant. A mixed model repeated measures ANCOVA using treatment, center, week, and treatment-by-week interaction in the model and baseline mean sleep score as the covariate; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -1.16, 95% CI 2-sided [-1.5 to -0.9]
Statistical Analysis 44: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.86, 95% CI 2-sided [-1.1 to -0.6]
Statistical Analysis 45: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < .0001, Mixed Model Repeated Measures ANCOVA; LS mean difference = -0.66, 95% CI 2-sided [-1.0 to -0.4]

5. Secondary Outcome: Percentage of Participants With Optimal Sleep Assessed Using MOS-SS
Description: Participant-rated 12 item questionnaire assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no), as well as a 9-item overall sleep problems index. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score minus lowest possible score divided by possible raw score range*100);total score range:0-100,higher score=more disturbance.
Time Frame: Baseline, Week 14
Population: FAS included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. Missing data were handled using LOCF method. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 182 | 182 | 175 | 182
Percentage of participants | 30.8 | 33.5 | 44.0 | 32.4
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P-values less than 0.05 (2-sided) considered statistically significant. Logistic regression method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.5370, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.71 to 1.95]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0109, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.16 to 3.18]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9613, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.61 to 1.68]

6. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS): Sub-scales at Week 14
Description: Participant-rated 12 item questionnaire assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no), as well as a 9-item overall sleep problems index. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score minus lowest possible score divided by possible raw score range*100);total score range:0-100,higher score=more intensity of attribute.
Time Frame: Baseline, Week 14
Population: FAS included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. Missing data were handled using LOCF method. 'N' (number of participants analyzed)=participants evaluable for this measure. 'n'=participants evaluable for specified category for each arm group.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 183 | 183 | 179 | 185
Units on a scale
  Sleep Disturbance (n=183,183,177,185) | -5.99 (1.79) | -13.18 (1.78) | -19.26 (1.84) | -18.70 (1.78)
  Snoring (n=172,174,174,177) | -0.03 (1.75) | 1.17 (1.73) | 4.89 (1.75) | 5.87 (1.73)
  Shortness of Breath, Headache (n=182,182,177,184) | -0.67 (1.92) | -9.62 (1.91) | -12.59 (1.96) | -9.91 (1.91)
  Quantity of Sleep (n=182,182,175,182) | 0.41 (0.10) | 0.61 (0.10) | 0.91 (0.11) | 0.76 (0.10)
  Sleep Adequacy (n=183,183,179,185) | 7.62 (1.93) | 10.19 (1.92) | 16.76 (1.96) | 11.97 (1.92)
  Somnolence (n=182,182,177,184) | -0.10 (1.50) | 0.67 (1.49) | 0.61 (1.53) | 1.92 (1.49)
  Overall Sleep Problem Index (n=181,181,174,184) | -4.83 (1.35) | -9.19 (1.34) | -13.07 (1.39) | -11.72 (1.34)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; Sleep Disturbance: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p < .0001, ANCOVA; LS mean difference = -12.71, 95% CI 2-sided [-17.56 to -7.86]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; LS mean difference = -13.28, 95% CI 2-sided [-18.18 to -8.38]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0038, ANCOVA; LS mean difference = -7.20, 95% CI 2-sided [-12.06 to -2.33]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 600 mg; Snoring: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0142, ANCOVA; LS mean difference = 5.90, 95% CI 2-sided [1.19 to 10.61]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0414, ANCOVA; LS mean difference = 4.92, 95% CI 2-sided [0.19 to 9.66]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.6165, ANCOVA; LS mean difference = 1.21, 95% CI 2-sided [-3.53 to 5.95]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 600 mg; Shortness of Breath, Headache: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0005, ANCOVA; LS mean difference = -9.24, 95% CI 2-sided [-14.44 to -4.05]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < .0001, ANCOVA; LS mean difference = -11.92, 95% CI [-17.17 to -6.68]
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.0008, ANCOVA; LS mean difference = -8.95, 95% CI 2-sided [-14.16 to -3.74]
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 600 mg; Quantity of Sleep: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0127, ANCOVA; LS mean difference = 0.36, 95% CI 2-sided [0.08 to 0.64]
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0005, ANCOVA; LS mean difference = 0.50, 95% CI 2-sided [0.22 to 0.79]
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 300 mg; Quality of Sleep: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.1453, ANCOVA; LS mean difference = 0.21, 95% CI 2-sided [-0.07 to 0.49]
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 600 mg; Sleep Adequacy: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.1033, ANCOVA; LS mean difference = 4.34, 95% CI 2-sided [-0.88 to 9.57]
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.0007, ANCOVA; LS mean difference = 9.14, 95% CI 2-sided [3.88 to 14.41]
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.3370, ANCOVA; LS mean difference = 2.56, 95% CI 2-sided [-2.68 to 7.81]
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 600 mg; Somnolence: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.3308, ANCOVA; LS mean difference = 2.01, 95% CI 2-sided [-2.05 to 6.07]
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.7364, ANCOVA; LS mean difference = 0.70, 95% CI 2-sided [-3.39 to 4.80]
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; p = 0.7132, ANCOVA; LS mean difference = 0.76, 95% CI 2-sided [-3.31 to 4.84]
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 600 mg; Overall sleep Problem Index: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0002, ANCOVA; LS mean difference = -6.90, 95% CI 2-sided [-10.54 to -3.25]
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p < .0001, ANCOVA; LS mean difference = -8.25, 95% CI 2-sided [-11.94 to -4.55]
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.0197, ANCOVA; LS mean difference = -4.36, 95% CI 2-sided [-8.02 to -0.70]

7. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Subscale Scores at Week 14
Description: FIQ: 20-item self-administered questionnaire designed to assess areas such as health status, progress, and outcomes in participants with fibromyalgia. 11 items related to physical functioning, other items assess pain, fatigue, stiffness, difficulty working, and symptoms of anxiousness and depression. FIQ contains 10 sub-scales scored from 0 to 10, with higher scores indicating more impairment in the subscale attribute. Total score range from 0 to 100 with higher scores indicating more impairment.
Time Frame: Baseline, Week 14
Population: FAS included all randomized participants who received at least 1 dose of study medication, regardless of medication compliance. Missing data were imputed using LOCF method. 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n'=participants evaluable for specified category for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 183 | 184 | 179 | 186
Units on a scale
  FIQ Physical Impairment (n=183,184,179,186) | -0.09 (0.14) | -0.26 (0.14) | -0.35 (0.14) | -0.26 (0.14)
  FIQ Feel Good (n=182,184,178,183) | -1.15 (0.22) | -1.11 (0.22) | -1.77 (0.22) | -1.26 (0.22)
  FIQ Work Missed (n=182,181,178,184) | -0.13 (0.19) | -0.29 (0.18) | -0.75 (0.19) | -0.27 (0.18)
  FIQ Do Work (n=182,183,179,185) | -0.90 (0.18) | -1.04 (0.18) | -1.60 (0.18) | -0.98 (0.18)
  FIQ Pain (n=183,184,179,185) | -0.97 (0.17) | -1.18 (0.17) | -1.72 (0.17) | -1.10 (0.17)
  FIQ Fatigue (n=183,184,179,184) | -0.81 (0.18) | -0.86 (0.18) | -1.36 (0.18) | -1.05 (0.18)
  FIQ Rested (n=183,184,179,185) | -0.94 (0.19) | -1.17 (0.19) | -1.47 (0.20) | -1.40 (0.19)
  FIQ Stiffness (n=183,184,179,185) | -1.06 (0.18) | -1.02 (0.18) | -1.28 (0.18) | -0.94 (0.18)
  FIQ Anxiety (n=183,184,179,185) | -0.48 (0.20) | -0.66 (0.20) | -1.12 (0.20) | -0.68 (0.20)
  FIQ Depression (n=181,184,179,184) | -0.22 (0.20) | -0.56 (0.20) | -1.19 (0.20) | -0.43 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; FIQ Physical Impairment: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.3627, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.54 to 0.20]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1686, ANCOVA; LS mean difference = -0.26, 95% CI 2-sided [-0.63 to 0.11]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3468, ANCOVA; LS mean difference = -0.18, 95% CI 2-sided [-0.55 to 0.19]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 600 mg; FIQ Feel Good: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.7147, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.71 to 0.49]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.0409, ANCOVA; LS mean difference = -0.63, 95% CI 2-sided [-1.23 to -0.03]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.9077, ANCOVA; LS mean difference = 0.04, 95% CI 2-sided [-0.56 to 0.63]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 600 mg; FIQ Work Missed: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.5923, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.64 to 0.37]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.0174, ANCOVA; LS mean difference = -0.61, 95% CI 2-sided [-1.12 to -0.11]
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.5408, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.66 to 0.35]
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 600 mg; FIQ Do Work: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.7236, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.57 to 0.40]
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.0045, ANCOVA; LS mean difference = -0.71, 95% CI 2-sided [-1.19 to -0.22]
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.5613, ANCOVA; LS mean difference = -0.14, 95% CI [-0.63 to 0.34]
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 600 mg; FIQ Pain: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.5609, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.60 to 0.33]
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p = 0.0016, ANCOVA; LS mean difference = -0.75, 95% CI 2-sided [-1.22 to -0.28]
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p = 0.3692, ANCOVA; LS mean difference = -0.21, 95% CI 2-sided [-0.68 to 0.25]
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 600 mg; FIQ Fatigue: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.3294, ANCOVA; LS mean difference = -0.24, 95% CI 2-sided [-0.73 to 0.25]
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.0270, ANCOVA; LS mean difference = -0.56, 95% CI 2-sided [-1.05 to -0.06]
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.8432, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.54 to 0.44]
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 600 mg; FIQ Rested: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0806, ANCOVA; LS mean difference = -0.46, 95% CI 2-sided [-0.98 to 0.06]
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; p = 0.0470, ANCOVA; LS mean difference = -0.53, 95% CI 2-sided [-1.06 to -0.01]
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 19]; Test type: Superiority or Other; p = 0.3845, ANCOVA; LS mean difference = -0.23, 95% CI 2-sided [-0.75 to 0.29]
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 600 mg; FIQ Stiffness: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.6326, ANCOVA; LS mean difference = 0.12, 95% CI 2-sided [-0.37 to 0.60]
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 22]; Test type: Superiority or Other; p = 0.3740, ANCOVA; LS mean difference = -0.22, 95% CI 2-sided [-0.71 to 0.27]
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 22]; Test type: Superiority or Other; p = 0.8936, ANCOVA; LS mean difference = 0.03, 95% CI 2-sided [-0.45 to 0.52]
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 600 mg; FIQ Anxiety: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.4743, ANCOVA; LS mean difference = -0.19, 95% CI 2-sided [-0.73 to 0.34]
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; p = 0.0192, ANCOVA; LS mean difference = -0.64, 95% CI 2-sided [-1.18 to -0.10]
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 25]; Test type: Superiority or Other; p = 0.5101, ANCOVA; LS mean difference = -0.18, 95% CI 2-sided [-0.71 to 0.35]
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 600 mg; FIQ Depression: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.4617, ANCOVA; LS mean difference = -0.20, 95% CI 2-sided [-0.75 to 0.34]
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 7, analysis 28]; Test type: Superiority or Other; p = 0.0006, ANCOVA; LS mean difference = -0.97, 95% CI 2-sided [-1.51 to -0.42]
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 7, analysis 28]; Test type: Superiority or Other; p = 0.2290, ANCOVA; LS mean difference = -0.33, 95% CI 2-sided [-0.88 to 0.21]

8. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Total Scores at Week 14
Description: as for outcome 7
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 179 | 186
Units on a scale | -6.94 (1.30) | -8.11 (1.29) | -12.79 (1.32) | -8.38 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.4200, ANCOVA; LS mean difference = -1.44, 95% CI 2-sided [-4.95 to 2.06]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0012, ANCOVA; LS mean difference = -5.85, 95% CI 2-sided [-9.38 to -2.31]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.5126, ANCOVA; LS mean difference = -1.17, 95% CI 2-sided [-4.68 to 2.34]

9. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Health Survey at Week 14
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; Physical Component Score and Mental Component Score. Total score range for the summary scores = 0- 100, where higher score represents higher level of functioning.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 178 | 186
Units on a scale
  Physical Functioning (n=184,184,177,186) | 4.64 (1.32) | 5.22 (1.31) | 6.63 (1.35) | 4.13 (1.31)
  Physical Role Limitations (n=183,183,177,185) | 4.01 (1.63) | 4.40 (1.62) | 5.50 (1.66) | 5.03 (1.62)
  Emotional Role Limitations (n=183,183,177,185) | -2.31 (1.94) | 1.44 (1.93) | 3.93 (1.98) | 1.56 (1.93)
  Social Functioning (n=183,184,178,186) | 0.75 (1.77) | 4.10 (1.76) | 5.76 (1.81) | 3.60 (1.76)
  Mental Health (n=183,184,178,186) | -1.67 (1.35) | 1.65 (1.34) | 4.25 (1.38) | 2.41 (1.34)
  Bodily Pain (n=183,184,178,186) | 4.95 (1.31) | 7.77 (1.30) | 10.32 (1.33) | 7.53 (1.30)
  Vitality (n=183,184,178,186) | 4.15 (1.42) | 4.89 (1.41) | 9.25 (1.45) | 7.29 (1.41)
  General Health Perception (n=183,184,177,186) | 0.94 (1.16) | 2.76 (1.15) | 3.67 (1.18) | 2.21 (1.14)
  Mental Component Score (n=182,183,176,184) | -1.27 (0.81) | 0.87 (0.81) | 2.39 (0.83) | 1.35 (0.81)
  Physical Component Score (n=182,183,176,184) | 2.47 (0.52) | 2.60 (0.52) | 3.01 (0.53) | 2.34 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; Physical functioning: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.7781, ANCOVA; LS mean difference = -0.51, 95% CI 2-sided [-4.07 to 3.05]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.2792, ANCOVA; LS mean difference = 1.99, 95% CI 2-sided [-1.62 to 5.59]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7512, ANCOVA; LS mean difference = 0.58, 95% CI 2-sided [-3.00 to 4.15]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 600 mg; Physical role Limitations: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.6490, ANCOVA; LS mean difference = 1.02, 95% CI 2-sided [-3.39 to 5.43]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.5105, ANCOVA; LS mean difference = 1.50, 95% CI 2-sided [-2.96 to 5.96]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.8625, ANCOVA; LS mean difference = 0.39, 95% CI 2-sided [-4.04 to 4.82]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 600 mg; Emotional Role Limitations: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.1489, ANCOVA; LS mean difference = 3.87, 95% CI 2-sided [-1.39 to 9.12]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.0213, ANCOVA; LS mean difference = 6.24, 95% CI 2-sided [0.93 to 11.54]
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.1620, ANCOVA; LS mean difference = 3.75, 95% CI 2-sided [-1.51 to 9.02]
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 600 mg; Social Functioning: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.2446, ANCOVA; LS mean difference = 2.85, 95% CI 2-sided [-1.95 to 7.65]
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.0429, ANCOVA; LS mean difference = 5.01, 95% CI 2-sided [0.16 to 9.85]
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.1721, ANCOVA; LS mean difference = 3.35, 95% CI 2-sided [-1.46 to 8.16]
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 600 mg; Mental Health: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0291, ANCOVA; LS mean difference = 4.08, 95% CI 2-sided [0.42 to 7.74]
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.0017, ANCOVA; LS mean difference = 5.93, 95% CI 2-sided [2.23 to 9.62]
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.0763, ANCOVA; LS mean difference = 3.32, 95% CI 2-sided [-0.35 to 6.99]
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 600 mg; Bodily Pain: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.1524, ANCOVA; LS mean difference = 2.58, 95% CI 2-sided [-0.95 to 6.11]
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.0032, ANCOVA; LS mean difference = 5.36, 95% CI 2-sided [1.80 to 8.93]
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.1180, ANCOVA; LS mean difference = 2.82, 95% CI 2-sided [-0.72 to 6.36]
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 600 mg; Vitality: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.1081, ANCOVA; LS mean difference = 3.15, 95% CI 2-sided [-0.69 to 6.99]
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.0101, ANCOVA; LS mean difference = 5.10, 95% CI 2-sided [1.22 to 8.99]
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.7031, ANCOVA; LS mean difference = 0.75, 95% CI 2-sided [-3.10 to 4.60]
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 600 mg; General Health Perception: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.4253, ANCOVA; LS mean difference = 1.27, 95% CI 2-sided [-1.86 to 4.39]
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 22]; Test type: Superiority or Other; p = 0.0910, ANCOVA; LS mean difference = 2.73, 95% CI 2-sided [-0.44 to 5.89]
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 22]; Test type: Superiority or Other; p = 0.2526, ANCOVA; LS mean difference = 1.82, 95% CI 2-sided [-1.30 to 4.95]
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 600 mg; Mental Component Score: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0195, ANCOVA; LS mean difference = 2.62, 95% CI 2-sided [0.42 to 4.82]
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p = 0.0013, ANCOVA; LS mean difference = 3.66, 95% CI 2-sided [1.44 to 5.88]
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p = 0.0568, ANCOVA; LS mean difference = 2.14, 95% CI 2-sided [-0.06 to 4.34]
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 600 mg; Physical Component Score: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.8529, ANCOVA; LS mean difference = -0.13, 95% CI 2-sided [-1.54 to 1.27]
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 9, analysis 28]; Test type: Superiority or Other; p = 0.4564, ANCOVA; LS mean difference = 0.54, 95% CI 2-sided [-0.88 to 1.96]
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 9, analysis 28]; Test type: Superiority or Other; p = 0.8576, ANCOVA; LS mean difference = 0.13, 95% CI 2-sided [-1.28 to 1.54]

10. Secondary Outcome: Change From Baseline in Multidimensional Assessment of Fatigue (MAF) at Week 14
Description: MAF is a 16-item self-administered questionnaire that yields a Global Fatigue Index (GFI), measures 4 dimensions of fatigue: degree and severity, amount of distress it causes, its timing and degree to which fatigue interferes with activities of daily living. Only 15 items are used to calculate the GFI. GFI score range from 1 (no fatigue) to 50 (severe fatigue).
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 183 | 176 | 175 | 181
Units on a scale | -1.91 (0.62) | -2.78 (0.63) | -3.32 (0.64) | -2.19 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.7384, ANCOVA; LS mean difference = -0.29, 95% CI 2-sided [-1.98 to 1.40]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.1044, ANCOVA; LS mean difference = -1.41, 95% CI 2-sided [-3.12 to 0.29]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.3137, ANCOVA; LS mean difference = -0.87, 95% CI 2-sided [-2.58 to 0.83]

11. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) at Week 14
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 182 | 181 | 176 | 185
Units on a scale
  HADS Anxiety (HADS-A) Total | -0.31 (0.25) | -0.42 (0.25) | -0.81 (0.26) | -0.90 (0.25)
  HADS Depression (HADS-D) Total | -0.11 (0.24) | -0.33 (0.24) | -0.70 (0.25) | 0.04 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; HADS-Anxiety Total: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.0900, ANCOVA; LS mean difference = -0.59, 95% CI 2-sided [-1.28 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1564, ANCOVA; LS mean difference = -0.50, 95% CI 2-sided [-1.20 to 0.19]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.7519, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.80 to 0.58]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 600 mg; HADS-Depression Total: P-values less than 0.05 (2-sided) considered statistically significant. ANCOVA method was used with treatment and center in the model, and the baseline score as covariate; Test type: Superiority or Other; p = 0.6416, ANCOVA; LS mean difference = 0.15, 95% CI 2-sided [-0.50 to 0.80]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.0778, ANCOVA; LS mean difference = -0.59, 95% CI 2-sided [-1.25 to 0.07]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.5191, ANCOVA; LS mean difference = -0.21, 95% CI 2-sided [-0.87 to 0.44]

12. Secondary Outcome: Change From Baseline in Pain Visual Analogue Scale (VAS) Scores at Week 14
Description: Pain visual analog scale (VAS): Participants assessed the severity of their pain using a 100 mm visual analog scale (VAS). The scale ranged from 0 (no pain) to 100 (worst possible pain), measurement on a scale corresponds to the magnitude of their pain.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 181 | 186
mm | -10.30 (1.67) | -12.86 (1.66) | -17.75 (1.69) | -11.74 (1.66)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.5340, ANCOVA; LS mean difference = -1.44, 95% CI 2-sided [-5.97 to 3.09]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0014, ANCOVA; LS mean difference = -7.44, 95% CI 2-sided [-12.00 to -2.88]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2694, ANCOVA; LS mean difference = -2.56, 95% CI 2-sided [-7.09 to 1.98]

13. Secondary Outcome: Total Daily Acetaminophen Dose
Description: Acetaminophen (up to 4 gram/day as needed for pain relief) was an allowable concomitant medication as a rescue therapy. The total daily acetaminophen dose taken during double-blind treatment was calculated for each participant as: (total acetaminophen dose during the study) divided by (total number of study days).
Time Frame: Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/day
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Number analyzed (Participants) | 184 | 184 | 182 | 186
mg/day | 460.65 (125.43) | 449.14 (124.79) | 508.53 (126.71) | 724.42 (124.72)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 600 mg; P-values less than 0.05 (2-sided) considered statistically significant. P value was calculated using analysis of variance (ANOVA), with treatment and center in the model; Test type: Superiority or Other; p = 0.1277, ANCOVA; LS mean difference = 263.77, 95% CI 2-sided [-75.78 to 603.33]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 450 mg; P-values less than 0.05 (2-sided) considered statistically significant. P value was calculated using ANOVA, with treatment and center in the model; Test type: Superiority or Other; p = 0.7829, ANCOVA; LS mean difference = 47.89, 95% CI 2-sided [-293.2 to 389.02]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.9471, ANCOVA; LS mean difference = -11.51, 95% CI 2-sided [-351.9 to 328.86]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Pregabalin 300 mg | Pregabalin 450 mg | Pregabalin 600 mg
Serious Adverse Events (participants affected / at risk) | 4/184 | 2/184 | 8/182 | 4/186
Other Adverse Events (participants affected / at risk) | 97/184 | 137/184 | 141/182 | 154/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | Pregabalin 300 mg (N=184) | Pregabalin 450 mg (N=182) | Pregabalin 600 mg (N=186)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Cerebrovascular accident (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | Pregabalin 300 mg (N=184) | Pregabalin 450 mg (N=182) | Pregabalin 600 mg (N=186)
Vertigo (Ear and labyrinth disorders) | 4 | 13 | 12 | 15
Vision blurred (Eye disorders) | 1 | 6 | 9 | 13
Constipation (Gastrointestinal disorders) | 8 | 18 | 12 | 15
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 4 | 16 | 20 | 20
Nausea (Gastrointestinal disorders) | 20 | 22 | 6 | 12
Fatigue (General disorders) | 15 | 14 | 26 | 17
Oedema peripheral (General disorders) | 7 | 19 | 15 | 27
Influenza (Infections and infestations) | 6 | 5 | 7 | 10
Nasopharyngitis (Infections and infestations) | 7 | 7 | 10 | 6
Weight increased (Investigations) | 6 | 24 | 24 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 6 | 5
Disturbance in attention (Nervous system disorders) | 4 | 10 | 12 | 15
Dizziness (Nervous system disorders) | 28 | 68 | 76 | 93
Headache (Nervous system disorders) | 30 | 27 | 25 | 16
Somnolence (Nervous system disorders) | 11 | 37 | 24 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.